CLINICAL TRIAL: NCT07142070
Title: Evaluation of the Effect of Systemic Retinoic Acid Use on Micro Ribonucleic Acid (mRNA) Expression in Saliva and Serum
Brief Title: Effect of Systemic Retinoic Acid Use on Micro Ribonucleic Acid (mRNA) Expression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melis Yilmaz, Assistant Prof Dr, Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1386
Record Dates: First submitted 2025-07-25; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Diseases; Inflammation
Keywords: periodontal disease; miRNA
MeSH Terms: conditions — Periodontal Diseases; Inflammation | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: Saliva, serum collected for analyzing tnf-a, miRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Salivary, serum, miRNA, TNF-a observation Saliva, serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for TNF-a using commercial ELISA kits (Elabscience, Houston, Texas, USA and Bioaasay Technology Laboratory (BT-Lab), Shanghai, China, respectively) according to the manufacturer's instructions.
  Interventions: Other: Saliva, serum sampling; Drug: oral isotretinoin

INTERVENTIONS:
Other: Saliva, serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant (Periopaper, Oraflow Inc., Plainview, NY, USA). Saliva, serum were then stored at -80 °C until analysis.
Drug: oral isotretinoin — oral isotretinoin

SUMMARY:
Ribonucleic acids (RNA) are molecules that transfer genetic information from the nucleus to the cytoplasm for protein translation. A subgroup of non-coding or non-messenger RNAs, known as microRNAs (miRNAs), regulates the expression of complementary mRNAs without coding for proteins. In this study, the investigators aimed to evaluate the effect of systemically administered oral isotretinoin on gingival health in terms of microRNA (miRNA), a molecule of interest in periodontal research, before, during, and after treatment.

DETAILED DESCRIPTION:
Healthy participants (n:25) enrolled for this study. Samples will be collected for each patient at the following time points: immediately before the initiation of retinoic acid treatment, during treatment at week 5 (T1), during treatment at month 5 (T2), and three months after the end of treatment (T3).

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* over 18 and under 45 years of age
* have at least 20 natural permanent teeth in occlusion excluding third molars,
* not be pregnant,
* have not used any antimicrobial and/or anti-inflammatory drugs in the past 3 months,
* have not received periodontal treatment in the past 6 months,
* have not undergone surgical periodontal treatment within the past year.

Exclusion Criteria:

* history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)
* nonsurgical periodontal treatment (previous 6 months)
* surgical periodontal treatment (previous 12 months)
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 6 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Saliva, serum samples processing and analyses | 1 month
  Saliva, serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for TNF-a using commercial ELISA kits. RT-qPCR-based miRNA gene expression analyses will be performed using Two-Step qRT-PCR Kits (Thermo Fisher Scientific, MA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No